CLINICAL TRIAL: NCT00857350
Title: The Prevalence of HIV Drug Resistance and Transmission Risk in Opioid Agonist Treatment
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, David Fiellin, Associate Professor of Medicine, Investigative Medicine and Public Health, Yale University
Other Study IDs: 0709003082
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: HIV Positive; Opioid Dependence; Opioid Agonist Treatment; HIV Infections
Keywords: HIV; resistance; opioid dependence
MeSH Terms: conditions — HIV Seropositivity; Opioid-Related Disorders; HIV Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV+, opiod dependent

SUMMARY:
HIV drug resistance presents a significant public heath problem. This proposal is designed to explore the association between ongoing illicit drug use and the prevalence of HIV drug resistance among HIV+ opioid dependent patients receiving opioid agonist treatment with the following hypotheses:

1. Hypothesis 1: The prevalence of HIV drug resistance will range between 10% and 30%.
2. Hypothesis 2: Patients with evidence of ongoing illicit drug use will be more likely to have HIV drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Opioid dependent
* Receiving methadone or buprenorphine for at least one month

Exclusion Criteria:

* age < 18 years
* current dementia;
* inability to read or understand English
* inability to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV+, opioid dependent
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
HIV drug resistance | Cross sectional

SECONDARY OUTCOMES:
Illicit drug use | 6 months
HIV transmission risk behaviors | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Fiellin, MD, Principal Investigator — Yale University; Jeanette Tetrault, MD, Principal Investigator — Yale University
Locations (1):
- Yale University Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Result] Tetrault JM, Kozal MJ, Chiarella J, Sullivan LE, Dinh AT, Fiellin DA. Association between risk behaviors and antiretroviral resistance in HIV-infected patients receiving opioid agonist treatment. J Addict Med. 2013 Mar-Apr;7(2):102-7. doi: 10.1097/ADM.0b013e31827f9bdf. PMID 23388678